CLINICAL TRIAL: NCT01169558
Title: First-Line Bevacizumab and Chemotherapy in Metastatic Cancer of the Colon or Rectum First BEAT (Bevacizumab Expanded Access Trial)- Brazilian Extension
Brief Title: A Study of Bevacizumab (Avastin) in Combination With Chemotherapy in Participants With Metastatic Cancer of the Colon or Rectum.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20552
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Results first posted 2016-10-18 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab will be administered in combination with fluoropyrimidine-based chemotherapy as first line treatment in participants with metastatic cancer of the colon or rectum until disease progression or study completion.
  Interventions: Drug: Bevacizumab; Drug: Fluoropyrimidine-based Chemotherapy

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg bevacizumab administered intravenously every 2 weeks or 7.5 mg/kg bevacizumab administered intravenously every 3 weeks according to the standard chemotherapy regimen.
  Other Names: Avastin
Drug: Fluoropyrimidine-based Chemotherapy — Fluoropyrimidine-based chemotherapy administered according to standard of care.

SUMMARY:
This expanded access study will assess the safety and efficacy of intravenous bevacizumab (5 mg/kg every 2 weeks or 7.5 mg/kg every 3 weeks) in combination with fluoropyrimidine-based chemotherapy as first line treatment in participants with metastatic cancer of the colon or rectum. The anticipated time on study treatment is 3-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated metastatic colon or rectal cancer;
* Scheduled to begin fluoropyrimidine-based chemotherapy as a first line treatment.

Exclusion Criteria:

* Prior chemotherapy for metastatic colon or rectal cancer;
* Planned radiotherapy for underlying disease;
* central nervous system metastases;
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days before study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (14):
- Brazil (14):
  - Belo Horizonte
  - Brasília
  - Campinas
  - Caxias do Sul
  - Curitiba
  - Fortaleza
  - Ijuí
  - João Pessoa
  - Porto Alegre
  - Recife
  - Ribeirão Preto
  - Rio de Janeiro
  - Salvador
  - São Paulo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 168 participants were enrolled in the study of which 162 received at least one dose of study drug. Only those who received at least one dose of study medication were included in the Intent to Treat (ITT) population, which is the population reported.
Groups:
- Bevacizumab: Bevacizumab (5 mg/kg intravenously every 2 weeks or 7.5 mg/kg intravenously every 3 weeks) was administered in combination with fluoropyrimidine-based chemotherapy as first line treatment in participants with metastatic cancer of the colon or rectum until disease progression or study completion.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 162
Completed | 6
Not Completed | 156
Not completed — Disease progression | 98
Not completed — Adverse Event | 25
Not completed — Withdrawal of Consent | 8
Not completed — Medical Decision | 7
Not completed — Stable Disease | 4
Not completed — Lost to Follow-up | 4
Not completed — Need for Surgery | 4
Not completed — Non-compliance | 2
Not completed — Protocol Violation | 2
Not completed — Partial response | 2

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population included all participants receiving at least one dose of the study drug.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 162
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (13.1)
Gender [Count of Participants; unit: Participants]
  Female | 89
  Male | 73

OUTCOME MEASURES:

1. Primary Outcome: Safety: Number of Participants With Serious and Specific Adverse Events
Description: A serious adverse event was defined as any experience that suggested a significant hazard, contraindication, side effect, or precaution, and fulfilled any of the following criteria: fatal (resulted in death), life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was medically significant or required intervention to prevent any of the other outcomes listed here. Specific adverse events (Spec AEs) included the following: hypertension, bleeding/hemorrhage, proteinuria, wound healing complications, thrombosis/thrombus/embolism (t/t/e), thrombosis/thrombus/embolism - vascular access, gastrointestinal perforation, and infusion (injection) site reaction.
Time Frame: Up to approximately 3 years
Population: The intent to treat (ITT) population included all participants receiving at least one dose of the study drug. This population was primarily used for the reporting of safety information.
Measure: Number; unit: participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 162
participants
  Serious Adverse Events | 50
  Spec AEs: Hypertension | 57
  Spec AEs: Bleeding/hemorrhage | 42
  Spec AEs: Proteinuria | 22
  Spec AEs:Wound healing complications | 6
  Spec AEs: Thrombosis/thrombus/embolism | 5
  Spec AEs: T/t/e - Vascular Access | 2
  Spec AEs: Gastrointestinal perforation | 2
  Spec AEs: Infusion (injection) Site Reaction | 2

2. Secondary Outcome: Efficacy: Overall Survival
Description: Overall survival was measured as the time from start of first bevacizumab administration to death. For participants who were alive at the end of the study, data on survival were censored at the time of the last contact. Reported is the median duration of overall survival.
Time Frame: Up to approximately 3 years
Population: 158 participants from the ITT population were included in the analysis. Four participants were excluded from the ITT population due to protocol deviation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 158
months | 21.6 [18.3 to 25.5]

3. Secondary Outcome: Efficacy: Time to Disease Progression
Description: Time to disease progression was measured as the time from start of first bevacizumab administration to investigator-assessed progression. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. For participants without disease progression at the end of the study, date and time to progression were censored at the last investigator assessment. Reported is the median time to disease progression.
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 158
months | 11.4 [9.5 to 13.9]

4. Secondary Outcome: Efficacy: Progression-free Survival
Description: Progression-free survival (PFS) was measured as the time from start of first bevacizumab administration to investigator-assessed progression or death, whichever occurred first. Progression was defined using RECIST v1.0, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Reported is the median time of PFS.
Time Frame: Up to approximately 3 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 158
months | 11.0 [9.5 to 13.9]

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Description: The intent to treat (ITT) population included all participants receiving at least one dose of the study drug. This population was used for the reporting of safety information.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 50/162
Other Adverse Events (participants affected / at risk) | 153/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=162)
Diarrhoea (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Anal fistula (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Intestinal fistula (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 3
Bone marrow failure (Blood and lymphatic system disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
Infection (Infections and infestations) | 2
Abdominal wall abscess (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Genitourinary tract infection (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 4
Cachexia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1
Pyrexia (General disorders) | 3
Mucosal inflammation (General disorders) | 2
Asthenia (General disorders) | 1
Disease progression (General disorders) | 1
Seizure (Nervous system disorders) | 2
Cerebrovascular accident (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal colic (Renal and urinary disorders) | 1
Vesical fistula (Renal and urinary disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Immunodeficiency (Immune system disorders) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Vaginal fistula (Reproductive system and breast disorders) | 1
Thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=162)
Diarrhoea (Gastrointestinal disorders) | 80
Nausea (Gastrointestinal disorders) | 75
Abdominal pain (Gastrointestinal disorders) | 51
Vomiting (Gastrointestinal disorders) | 48
Stomatitis (Gastrointestinal disorders) | 42
Constipation (Gastrointestinal disorders) | 18
Rectal haemorrhage (Gastrointestinal disorders) | 9
Fatigue (General disorders) | 65
Pyrexia (General disorders) | 24
Influenza like illness (General disorders) | 11
Oedema peripheral (General disorders) | 9
Hypertension (Vascular disorders) | 57
Peripheral sensory neuropathy (Nervous system disorders) | 42
Headache (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 12
Proteinuria (Renal and urinary disorders) | 48
Decreased appetite (Metabolism and nutrition disorders) | 39
Dehydration (Metabolism and nutrition disorders) | 13
Rash (Skin and subcutaneous tissue disorders) | 28
Alopecia (Skin and subcutaneous tissue disorders) | 19
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15
Weight decreased (Investigations) | 19
Weight increased (Investigations) | 13
Upper respiratory tract infection (Infections and infestations) | 12
Depression (Psychiatric disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.